CLINICAL TRIAL: NCT03553030
Title: Early Insurgence of Coronary Artery Dysfunction in Prediabetic Patients With Monovessel Non Obstructive Coronary Stenosis May Condition Major Adverse Cardiac Events at 24 Months of Follow up.
Brief Title: Prediabetes and Non Obstructive Coronary Atherosclerosis.
Status: Completed | Type: Observational
Sponsor: University of Campania Luigi Vanvitelli (Other)
Responsible Party: Principal Investigator, Celestino Sardu, Principal investigator, University of Campania Luigi Vanvitelli
Other Study IDs: SecondUNI28.5.2018
Record Dates: First submitted 2018-05-29; First posted 2018-06-12 (Actual); Last update posted 2018-06-12 (Actual); Status verified 2018-06

CONDITIONS: PreDiabetes
MeSH Terms: conditions — Prediabetic State

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- prediabetics: patients with diagnosed of prediabetes.
  Interventions: Device: coronary artery angiography
- normo glycemics (controls): patients without diagnosed of prediabetes.
  Interventions: Device: coronary artery angiography

INTERVENTIONS:
Device: coronary artery angiography — In all patients authors performed a coronary artery angiography for detection of coronary artery stenosis.

SUMMARY:
Objectives: Prediabetes may condition an early endothelium dysfunction, and the development of non obstructive coronary stenosis (NOCS). Indeed, authors' study aim was to investigate the endothelial dysfunction, and Major Adverse Cardiac Events (MACE) in prediabetics vs. normo glycemic subjects.

Materials and Methods: 308 patients with evidence of left anterior descending (LAD) coronary NOCS (<50% luminal stenosis), will entere prospectively into a database. After assessment of endothelial coronary dysfunction by acetilcoline infusion, 86 propensity score matched (PSM) prediabetics and 86 PSM normoglycemics will be consecutive enrolled in the study.

DETAILED DESCRIPTION:
INTRODUCTION Prediabetes is a heterogeneous pathological condition diagnosed by the evidence of fasting plasma glucose of ≥5.6 mmol/L but <7.0 mmol/L (100-125 mg/dL; impaired fasting glucose [IFG]), a 2-hour glucose of ≥7.8 mmol/L but <11.1 mmol/L during a 75 g oral glucose tolerance test (GTT) (140-199 mg/dL; impaired glucose tolerance [IGT]), or a plasma hemoglobin (Hb) A1c of ≥5.7% but <6.5%. Epidemiological data confirm prediabetes as an increasing disease with a prevalence in the adults population of United States >38%. However, prediabetics present an increased risk to develop diabetes, and cardiovascular disease, then associated to worse prognosis. The common pathogenic mechanism linking prediabetes to cardiovascular disease is represented by the early insurgence of coronary artery dysfunction. It looks intuitive to speculate that, in prediabetics the hyperglycemia may early condition the coronary artery dysfunction, by a hyper activation of inflammatory and oxidative processes at level of endothelium covering the intima surface of coronary vessels. To date, the coronary artery dysfunction in prediabetics is well characterized by the endothelium dysfunction hyperglycemia induced. In fact, the endothelial dysfunction in prediabetics is characterized by a loss of vasodilation in response to sheer stress induced by release of an occlusive cuff (flow-mediated dilation) or pharmacological stimuli causing nitric oxide (NO) synthase activation such as acetylcholine. Moreover, in prediabetics the hyperglycemia may induce endothelial dysfunction evident in the early pathogenesis of atherosclerosis, such as it may be for patients with non obstructive coronary stenosis (NOCS). However, this early insurgence of coronary artery dysfunction in prediabetics may secondary lead to worse prognosis by an increasing number of Major Adverse Cardiac Events (MACE). On the other hand, actually a great discordance in literature exists about the correlation between NOCS in prediabetics and the associated clinical outcomes. In fact, authors recently reported that, asymptomatic prediabetics enrolled for early detection of coronary artery disease, and assessed by coronary computed tomography angiography, were not associated with an increased risk of subclinical coronary atherosclerosis. On the contrary, because the hyperglycemia may induce in prediabetics a higher expression of inflammatory and oxidative pathways, these multiple altered molecular pathways may consequently condition an endothelial dysfunction. However, limited data are actually evident about the impact of the glycemic status on the risk of subclinical coronary atherosclerosis in NOCS prediabetics as compared to normoglycemics patients. Therefore, author study hypothesis will be as first that, NOCS prediabetics vs. normoglycemics may present a higher level of inflammatory and oxidative markers. As second, these altered pathways may lead to an early endothelial dysfunction also in presence of monovessel NOCS. Finally, this pathogenic status may subsequently condition the worse prognosis in prediabetics vs. normoglycemics. Indeed, authors' study aim will be to investigate the endothelial dysfunction and the related MACE at 24 months of follow up in prediabetics vs. normo glycemic subjects with diagnosis of monovessel NOCS diagnosed by coronary angiography and infusion of acetylcholine.

METHODS Authors will screen at the Department of Cardiology, Hospital Cardarelli, Naples, Italy, and at Department of Cardiovascular Diseases, John Paul II Research and Care Foundation, Campobasso, Italy, patients having stable angina pectoris, with a positive stress test for myocardial ischemia, and no change in the frequency, duration, or intensity of clinical symptoms within 4 weeks, and referred for coronary artery angiography. However, these patients will receive a coronary angiography, and 267 patients with evidence of left anterior descending (LAD) coronary NOCS (<50% luminal stenosis), and no physiologically significant fractional flow reserve (FFR >0.80), will enter prospectively into a database. After the diagnosis of monovessel LAD-NOCS, authors will evaluate in these patients the endothelial coronary vascular function at baseline and after each infusion of acetylcholine. However these patients will be divided in subjects with normal endothelial function vs. subjects with endothelial dysfunction. Patients with no coronary disease detected by coronary angiography, presence of both obstructive and non-obstructive stenosis, left ventricular ejection fraction <50%, previous myocardial infarction, previous percutaneous coronary intervention and/or coronary bypass grafting, Tako-tsubo cardiomyopathy, myocarditis, impaired renal function or stroke will be excluded. To date 86 propensity score matched (PSM) prediabetics and 86 PSM normoglycemics will be consecutive enrolled in the study. Prediabetes will be defined by IFG, and IGT with an HbA1c value in the range of 6.4% (1). The analyses of all angiographic data will be performed by the interventional cardiologists, blinded to patient categorization, who will review selected cases with NOCS. After an overnight fast, plasma glucose and glycated haemoglobin (HbA1c) levels will be measured using enzymatic assays. At the Department of Medical, Surgical, Neurological, Aging and Metabolic Sciences, University of Campania "Luigi Vanvitelli", Italy, authors will practice for all patients quarterly clinical evaluation, routine analyses, plasma glucose and glycated haemoglobin (HbA1c) levels measurements, and cardiovascular evaluation as outpatients for 24 months after the coronarography. The study endpoints will be the assessment of oxidative stress, inflammatory tone, and MACE at 24 months follow up. The study will be conducted in accordance with the Declaration of Helsinki. The ethics committees of all participating institutions will approve the protocol. All patients will be informed about the study nature, and will give their written informed and signed consent to participate in the study.

Coronary angiography and endothelial function assessment. Experienced physician will perform routine diagnostic coronary angiography (General Electric, Discovery IGS 740) by using standard clinical protocols. Coronary angiography will be performed to discriminate and select patients with monovessel LAD and NOCS, as a stenosis <50% of vessel lumen, and with a fractionated flow reserve (FFr) >0.80 (8, 9). After the diagnosis of monovessel LAD-NOCS, in these patients authors will evaluate the endothelial coronary vascular function at baseline and after each infusion of acetylcholine. However, coronary artery diameter will be measured at baseline and after the infusion of acetylcholine by an independent investigator blinded to Doppler velocity data, and using a previously described computer-based image analysis system. The infusion protocol of acetylcholine will be terminated when the highest molar concentration of acetylcholine (1,024 mol/l) will be reached (8). Endothelial-dependent coronary blood flow (CBF) will be then calculated by the formula: CBF ¼ p(average peak velocity)(coronary artery diameter/2)2 (8). The inter observer and intra observer reproducibility of the CBF calculation will be about 5%. The maximal percent increase in CBF in response to acetylcholine compared with the CBF at baseline will be then calculated, and all measurements will be performed in the segment 5 mm distal to the tip of the Doppler guidewire. Moreover, after each acetylcholine infusion, the coronary artery diameter will be measured in the same segment of the vessel. The maximal effect of acetylcholine will be expressed as percent change in coronary artery diameter using quantitative coronary angiography (QCA, Medis Corporation, Leiden, the Netherlands) (representing epicardial endothelial function) and percent change in the CBF (representing microvascular endothelial function) relative to baseline (8).

Biochemical analyses. Venous blood samples, obtained from all participants in the study at baseline and during follow up phases, will be centrifuged at 3,000 rotations/min, and serum/plasma samples will be collected and stored at -80°C until assayed. Serum levels of high-sensitivity C-reactive protein (hs-CRP), Interleukine 1 (IL1) and 6 (IL 6), and TNF alpha will be measured as an inflammatory biomarker. In addition authors will measure the number of white blood cells (WBC), granulocytes, platelets, and blood values of Nitrotirosine as markers of oxidative stress on admission before coronary angiography and at follow up.

Statystical analysis SPSS version 23.0 (IBM statistics) will be used for all statistical analyses. Categorical variables will be presented as frequencies (percentages), and continuous variables as mean ± standard deviation. For comparisons between prediabetics and normoglycemics (controls) with normal epicardial endothelial function and those with epicardial endothelial dysfunction, propensity score matching will be developed from the predicted probabilities of a multivariable logistic regression model predicting mortality and events according to age, sex, hypertension, dyslipidaemia, smoking history, family history, baseline therapies, metabolic characteristics and coronary lesions. Overall survival and event-free survival will bee presented using Kaplan-Meier survival curves, and compared using the log-rank test. Univariable Cox models will be then used to compare event risks. The resulting hazard ratios (HRs) and 95% confidence intervals (CIs) will be reported. Two-tailed P values <.05 will be taken to indicate statistical significance.

ELIGIBILITY:
Inclusion Criteria:

* aged > 18 years.
* aged < 75 years.
* monovessel non obstructive coronary stenosis (as stenosis <50% of coronary artery lumen)

Exclusion Criteria:

* acute coronary syndrome,
* presence of of both obstructive and non-obstructive stenosis,
* left ventricular ejection fraction <50%,
* previous myocardial infarction,
* previous percutaneous coronary intervention and/or coronary bypass grafting,
* Tako-tsubo cardiomyopathy,
* myocarditis,
* impaired renal function
* stroke

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: a cohort of patients divided in prediabetics (n 86) vs. normoglycemics (n 86) that underwent coronary artery angiography for chest pain.
Sampling Method: Probability Sample
Enrollment: 172 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2017-07-01 (Actual); Study Completion 2018-01-01 (Actual)

PRIMARY OUTCOMES:
Major Adverse Cardiac Events (MACE). | 24 months.
  Authors will investigate the MACE, as post procedural and follow up angina, stroke, myocardial infarction, and re-hospitalization for acute coronary syndrome.

CONTACTS AND LOCATIONS:
Locations (1):
- Raffaele Marfella, Naples, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Sardu C, Paolisso P, Sacra C, Mauro C, Minicucci F, Portoghese M, Rizzo MR, Barbieri M, Sasso FC, D'Onofrio N, Balestrieri ML, Calabro P, Paolisso G, Marfella R. Effects of Metformin Therapy on Coronary Endothelial Dysfunction in Patients With Prediabetes With Stable Angina and Nonobstructive Coronary Artery Stenosis: The CODYCE Multicenter Prospective Study. Diabetes Care. 2019 Oct;42(10):1946-1955. doi: 10.2337/dc18-2356. Epub 2019 Feb 22. PMID 30796109